CLINICAL TRIAL: NCT00161694
Title: Effectiveness of an Oral Sucrose Solution in Reducing Pain and Anxiety Associated With Neonatal Ophthalmologic Examination
Brief Title: Use of Sucrose to Relieve Pain During Eye Exams in Infants
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: results did not show intervention was beneficial
Sponsor: Weill Medical College of Cornell University (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 0412007634
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2008-06-04 (Estimated); Status verified 2008-06

CONDITIONS: Apnea of Prematurity; Retinopathy of Prematurity; Pain
Keywords: pain control
MeSH Terms: conditions — Apnea; Retinopathy of Prematurity; Pain; Agnosia | interventions — sodium lactobionate sucrose solution

INTERVENTIONS:
Dietary Supplement: sucrose solution

SUMMARY:
The purpose of this study is to see if an oral sucrose solution can comfort premature infants during their necessary eye exams. The investigators believe that the use of this solution prior to the eye exams will lead to a decrease in pain as measured by a rise in heart rate and a fall in oxygen saturation. In addition this will lead to a decrease in events in the 12 hours following examination. Events include episodes when the infants temporarily stop breathing, have a drop in their heart rates, or have a drop in their oxygen levels.

ELIGIBILITY:
Inclusion Criteria:

* All premature infants admitted to the Neonatal Intensive Care Unit requiring serial dilated examinations to assess for retinopathy of prematurity will be candidates for this study. This includes all infants with a birthweight of less than 1500 g and infants between 1500 g and 2000 g who require supplemental oxygen.

Exclusion Criteria:

* Any infant who is unable to safely suckle 0.5 cc of fluid will be excluded from the study. This includes infants that are being maintained on ventilators and those with serious gastrointestinal complications that may be exacerbated by an oral fluid bolus.
* Any infant being maintained on narcotics for any reason will not be eligible for the study.
* All infants with major congenital anomalies will be excluded.

Min Age: 5 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2005-07

CONTACTS AND LOCATIONS:
Overall Officials: Tamara L Rousseau, MD, Principal Investigator — Neonatology Fellow at NYPH-Weill Cornell Medical Center
Locations (1):
- NYPH - Weill Cornell Medical Center, New York, New York, United States

REFERENCES:
- [Background] 1 American Academy of Pediatrics: screening Examination of Premature Infants for Retinopathy of Prematurity. Pediatrics 2001;108:809-811. 2 Laws DE,C Morton, MWeindling, D Clark. Systemic effects of screening for retinopathy of prematurity. Br J Opthalmol 1996;80:425-428. 3 Kumar H, S Naniwal, USingha, E Azad, VK Paul. Stress induced by screening for retinopathy of prematurity. J Pediatr Opthalmology and Strabismus. 2002;39:349-350. 4 Aguirre Rodriguez FJ, A Bonilla Perales, J Diez-Delgado Rubio, M Gonzales-Ripoll Garzon, J Arcos Martinez, J Lopez Munoz. An Pediatr (Barc) 2003;58:504-505. 5 Slevin M, JFA Murphy, L Daly, m o'Keefe. Retinopathy of prematurity screening, stress related response, the role of nesting. Br J Opthalmol 1997;81:762-764. 6 Als H, G Lawhon, E Brown et al. Individualized behavior and environmental care for the VLBW preterm infant at high risk for BPD: NICU and developmental outcome. Pediatrics 1986;78:1123-1132. 7 Stevens B, J Yamada, A Ohlsson. Sucrose for analgesia in newborn infants undergoing painful procedures (Cochrane Review). In The Cochrane Library, Issue 1, 2004. 8 Benis MM. Efficacy of sucrose analgesia for procedural pain in neonates. Dv Neonatal Care. 2002;2:93-100. 9 Masters-Harte LD. Sucrose analgesia for minor procedures in newborn infants. Ann Pharmacother 2001;35:947-952. 10 Akman I, EOzek, H Bilgen, T Ozgodan, D Cebeci. Sweet solutions and pacifiers for pain relief in newborn infants. The Journal of Pain 2002:3. 11 Blass EM. Behavioral and physiological consequences of suckling in rat and human newborns. Acta Paediatr Suppl 1994;397:71-76. 12 Campos RG. Soothing pain-elicited distress in infants with swaddling and pacifiers. Child Dev 1989;60:781-792. 13 Blass EM. Suckling and sucrose-induced analgesia in human newborns. Pain 1999;83:611-623. 14 Carbajal R, R Lenclen, V Gadjos, M Jugic, A Paupe. Crossover trial of analgesic efficacy of glucose and pacifier in very preterm neonates during subcutaneous injections. Pediatrics 2002;110:389-393. 15 Blass EM. Milk induced hypoalgesia in human newborns. Pediatrics 1997;99:825-829. 16 Carbajal R, S Veerapen, S Coulder, M Jugie, Y Ville. Analgesic effect of breast-feeding in term neonates: randomized controlled trial. British Medical Journal 2003;326:13. 17 Guala A. Glucose or sucrose as an analgesic for newborns: a randomized controlled blind trial. Minerva Pediatr 2001;53:271-274. 18 Anseloni VC. Age-dependency of analgesia elicited by intraoral sucrose in acute and persistent pain models. Pain 2002;97:93-103. 19 Willis D, J Chabot, I Radde, G Chance. Unsuspected hyperosmolality of oral solutions contributing to necrotizing enterocolitis in very-low-birth-weight infants. Pediatrics 1997;60:535-538. 20 American Academy of Pediatrics. Prevention and Management of Pain and Stress in the Neonate. Pediatrics 2000;105:454-461. 21 Morison S, R Grunau, T Oberlander, F Tim, M Whitfield. Relations between behavioral and cardiac autonomic reactivity to acute pain in preterm neonates. Clinical Journal of Pain 2001;17:350-358.